CLINICAL TRIAL: NCT04747457
Title: Development of Predictive Indicators of Homogeneous Propagation of Ultrasound and Elastic Waves During VCTE Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M138
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Liver Fibrosis
Keywords: FibroScan; Vibration Control Transient Elastography; Vibration Guided Transient Elastography; Liver Stiffness Measurement; VCTE; VGTE
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults and pediatric patients, all etiologies combined (Experimental)
  Interventions: Device: Research FibroScan

INTERVENTIONS:
Device: Research FibroScan — After having obtained the patient's Informed Consent Form signature, the following 3 examinations will be done:
  1. Standard examination [Reference CE-marked FibroScan]: the operator will need to find an optimal measurement area, and perform 10 valid measurements.
  2. Standard examination [Research FibroScan]: the operator must take 15 valid measurements at the same measurement point as the one used for the examination with the Reference FibroScan.
  3. Exploratory examination [Research FibroScan]: the operator needs to perform15 invalid measurements to acquire data in non-optimal regions of measurement (lungs, vessels, intestines, ribs, edges of the liver).

SUMMARY:
This is an European, prospective, interventional, and multicenter exploratory clinical investigation that will take place in 6 French sites and 200 patients will be included (adults and children). The study objective is to develop predictive indicators of homogeneous propagation of ultrasound and elastic waves to define an optimal region of interest for the measurement of liver stiffness during VCTE examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients, all etiologies combined
* Patient must be able to give written informed consent, or the parents in the case of a minor patient
* Patient affiliated to a social security system

Exclusion Criteria:

* Vulnerable patient- other than pediatric patients
* Pregnant or breastfeeding woman

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Validity criteria of the Liver Stiffness Measurement (LSM) by Vibration Controlled Transient Elastography (VCTE) (automatically assessed by the Reference and the Research FibroScan) | 7 months
  The validity criteria is an analysis of the measurement, automatically computed by the FibroScan. A measurement analyzed as "valid" leads to a reliable LSM whereas a measurement analyzed as "invalid" leads to a non-reliable LSM.

SECONDARY OUTCOMES:
The bias between the CAPc measured with the VCTE (Reference FibroScan) and the CAPc measured by the Vibration Guided Transient Elastography (VGTE) (Research FibroScan). | 7 months
Calculate the bias between the PCD measured by the VCTE (Reference FibroScan) and the PCD measured by the VGTE (Research FibroScan). | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Boursier, Pr, Principal Investigator — University Hospital, Angers
Locations (6):
- France (6):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Lille, Lille
  - Hôpital Saint Eloi, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice